CLINICAL TRIAL: NCT03566719
Title: Effectiveness of an Exercise Program for Prevention of Risk of Fall in a Community Dwelling Adults Over 55 Years
Brief Title: Effect of an Exercise Program on Risk of Fall in a Community Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Lúcia Morgado Martins (Other)
Responsible Party: Sponsor-Investigator, Sara Lúcia Morgado Martins, MSc, Escola Superior de Tecnologia da Saúde de Coimbra
Organization: Escola Superior de Tecnologia da Saúde de Coimbra (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: hdl.handle.net/10400.26/22351
Record Dates: First submitted 2018-04-18; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Elderly; Fall Risk; Fall
Keywords: Prevention; Active Ageing; Fall; Fall Risk; Exercise Programs
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: Exercise program
- Control group (No Intervention)

INTERVENTIONS:
Other: Exercise program — Intervention group has been submitted to an exercise program directed to prevent and reduce fall risk
  Arms: Intervention group

SUMMARY:
Background: Falls are a problem among the elderly population, it is known that currently about 30% of people over 65 years falls every year. The European Union estimates a cost of € 281 per inhabitant per year and a cost of € 25 billion per year for health care1 which translates into a significant economic impact. The World Health Organization2 argues that it is possible to reduce these costs through prevention and health promotion strategies. For this, it is important to raise awareness, evaluate risk factors and identify and implement intervention programs. Objective: To test the effect of an exercise program on the prevention of risk of fall. Methods: This study, which lasted 4 months, was experimental, prospective. The experimental group (EG) performed an exercise program and the control group (CG) maintained their usual routine. For the measurement and evaluation of the variables under study, were used: sociodemographic data questionnaire, self-efficacy for exercise scale, Portuguese version of the falls efficacy scale (FES), 10m walking speed (WS), Timed Up & Go test (TUG), step test and Hercules® Force Platform (static balance). A significance level of 5% (p ≤ 0.05) was considered for all comparisons.

ELIGIBILITY:
Inclusion Criteria:

* age equal or superior to 55
* community dwelling individuals

Exclusion Criteria:

* comprehension deficit
* significative heart disease
* restrictive breath disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Force Platform at 4 months | 0 and 4 months
  Static balance
Change from baseline Timed Up&Go at 4 months | 0 and 4 months
  Dynamic balance
Change from baseline Step test at 4 months | 0 and 4 months
  Muscular strength, motor coordination e inferior limb's agility
Change from baseline 10-meters walking test at 4 months | 0 and 4 months
  Walking speed
Change from baseline FES at 4 months | 0 and 4 months
  Fear of falling related by individuals and by their Daily live activity's execution
Change from baseline Self efficacy for exercise at 4 months | 0 and 4 months
  Self efficacy for exercise
Change from baseline Exercise program adherence at 4 months | 0 and 4 months
  Exercise program adherence 8number of sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Anabela C Martins, PhD, Study Chair — IPC ESTeSC Coimbra Health School

IPD SHARING:
Plan to Share IPD: Yes